CLINICAL TRIAL: NCT06020898
Title: Sodium Valproate in Patients With Acute Ischemic Stroke: a Pilot Randomized Trial
Brief Title: Sodium Valproate in Patients With Acute Ischemic Stroke
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Peiying Li, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LY2023-138-A
Record Dates: First submitted 2023-08-14; First posted 2023-09-01 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Sodium valproate; Acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Valproic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium valproate group (Experimental): Within 3 days after admission, 20mg/kg sodium valproate will be given daily. Specifically, 400mg sodium valproate will be infused within 5 minutes, followed by intravenous drip with 1mg/kg/h.
  Interventions: Drug: Sodium valproate
- Placebo group (Placebo Comparator): Within 3 days after admission, normal saline will be given daily in the same way.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Sodium valproate — Patients with acute ischemic stroke included in the study are randomly assigned to low-dose sodium valproate group, high-dose sodium valproate group and placebo group. Besides receiving conventional treatment for stroke, 10mg/kg sodium valproate, 20mg/kg sodium valproate or normal saline were given intravenously for 3 consecutive days, respectively.
  Arms: Sodium valproate group
Drug: Normal saline — Patients with acute ischemic stroke included in the study are randomly assigned to low-dose sodium valproate group, high-dose sodium valproate group and placebo group. Besides receiving conventional treatment for stroke, 10mg/kg sodium valproate, 20mg/kg sodium valproate or normal saline were given intravenously for 3 consecutive days, respectively.
  Arms: Placebo group

SUMMARY:
The purpose of this pilot trial is to investigate the feasibility, safety, and efficacy of sodium valproate in patients with acute ischemic stroke, and also explore the mechanism: whether valproate increases peripheral anti-inflammatory CD177+ neutrophil levels.

DETAILED DESCRIPTION:
Ischemic stroke is one of the leading causes of disability and mortality worldwide, which imposes a huge burden on families and society. Currently, the effective treatment strategies of ischemic stroke are limited. It is of great clinical value and significance to explore effective neuroprotective medications besides reperfusion therapy.

Sodium valproate is widely used in clinical practice, and its safety and tolerability has been confirmed. It is mainly used in the treatment of epilepsy, bipolar disorder, neuropathic pain and other diseases. In recent years, a number of preclinical studies have found that valproic acid has a potential neuroprotective effect in acute ischemic brain injury, which can decrease infarct volume, reduce blood-brain barrier damage, and improve neurological function. However, the neuroprotective mechanism of sodium valproate has not been fully revealed, and there is still a lack of clinical studies to clarify the neuroprotective effect of sodium valproate in patients with ischemic stroke.

The goal of this study is to test whether sodium valproate could become a new therapeutic approach for ischemic stroke. This prospective pilot study is intended to investigate the feasibility, safety, and efficacy of sodium valproate in patients with acute ischemic stroke, thus support the estimate of sample size for a future full trial. In addition, we will test the hypotheses that valproate increases peripheral anti-inflammatory CD177+ neutrophil levels.

Patients with acute ischemic stroke included in the study will be randomly assigned to sodium valproate group (20 mg/kg/d) or saline placebo group. Treatment will be started within 24 hours after stroke onset. The trial drug will be given intravenously for 3 consecutive days. The investigators evaluate whether sodium valproate can improve clinical outcomes and increase peripheral CD177+ neutrophil levels.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤age<75 years;
2. Admitted to hospital within 24 hours after the onset of neurological impairment symptoms consequent to acute ischemic stroke diagnosed by CT or MRI;
3. Not suitable for thrombolysis and mechanical thrombectomy;
4. Written informed consent.

Exclusion Criteria:

1. mRS ≥ 2 before the disease onset;
2. Refractory hypertension (SBP>180mmHg or DBP>110mmHg after antihypertensive treatment);
3. History of cerebral hemorrhage, intracranial tumor, cerebral arteriovenous malformation and aneurysm;
4. History of brain trauma, intracranial or spinal surgery within 3 months, major surgery or severe physical trauma within 1 month;
5. Signs of infection at time of admission;
6. History of malignancy or active autoimmune disease;
7. Use of glucocorticoids or other immunosuppressive medications;
8. Contraindications to sodium valproate: pregnancy; liver disease or severe hepatic insufficiency (ALT, AST 3 times higher than the upper normal limit); hemorrhagic risk (such as platelet count <100x109/L, APTT≥35s); allergy to sodium valproate, sodium divalproate, or valproamide; hepatic porphyria; combined use of mefloquine; mitochondrial diseases related to POLG mutations; known disorders of the urea cycle;
9. Use of medications containing active ingredients that can be converted to valproic acid, including sodium divalproate and valproamide;
10. Contraindications or intolerance for CT perfusion imaging;
11. Participating in other conflicting clinical trials;
12. Any other condition that investigators consider unsuitable such as mental illness, cognitive impairment, or inability to follow trial procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Favorable outcome at 90 days (the Modified Rankin Scale (mRS) score≤2) | Day 90
  The proportion of patients with favorable outcome, which is defined as the Modified Rankin Scale (mRS) score 0-2.

SECONDARY OUTCOMES:
Favorable outcome at 30 days (the Modified Rankin Scale (mRS) score≤2) | Day 30
  The proportion of patients with favorable outcome, which is defined as the Modified Rankin Scale (mRS) score 0-2.
NIH Stroke Scale (NIHSS) score at 3 days | Day 3
  The NIH Stroke Scale (NIHSS) score ranges from 0 to 42, where high scores mean a worse outcome.
NIH Stroke Scale (NIHSS) score at 7 days | Day 7
  The NIH Stroke Scale (NIHSS) score ranges from 0 to 42, where high scores mean a worse outcome.
Changes of lesion volume from baseline to day 7 | Day 7
  The infarct lesion volume will be measures on magnetic resonance imaging DWI and FLAIR.

OTHER OUTCOMES:
The peripheral CD177+ neutrophil levels | Day 3 and Day 7
  The CD177+ neutrophil levels in peripheral blood will be evaluated using flow cytometry.
The levels of inflammatory cytokines in peripheral blood | Day 3 and Day 7
  IL-1β、IL-2、IL-4、IL-5、IL-6、IL-8、IL-10、IL-12、IL-17A、IFN-α、IFN-γ、TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Peiying Li, Doctor, Principal Investigator — RenJi Hospital; Jieqing Wan, Doctor, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China